CLINICAL TRIAL: NCT03282786
Title: Comparison of Carbon Dioxide (CO2) to Air Insufflation in Colonoscopy in Patients With Inflammatory Bowel Disease
Acronym: CO2-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017-191-f-S
Record Dates: First submitted 2017-09-05; First posted 2017-09-14 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Carbon Dioxide (CO2); Colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CD patient with CO2 insufflation (Active Comparator): The investigators aim to include 76 Crohn's disease (CD) patients undergoing colonoscopy in whom CO2 insufflation during endoscopy should be used.
  Interventions: Other: carbon dioxide insufflation during colonoscopy
- CD patient with air insufflation (No Intervention): The investigators aim to include 76 Crohn's disease patients undergoing colonoscopy in whom air insufflation during endoscopy should be used.
- UC patient with CO2 insufflation (Active Comparator): The investigators aim to include 76 ulcerative colitis patients (UC) undergoing colonoscopy in whom CO2 insufflation during endoscopy should be used.
  Interventions: Other: carbon dioxide insufflation during colonoscopy
- UC patient with air insufflation (No Intervention): The investigators aim to include 76 ulcerative colitis patients undergoing colonoscopy in whom air insufflation during endoscopy should be used.

INTERVENTIONS:
Other: carbon dioxide insufflation during colonoscopy — Use of Carbon dioxide instead of air insufflation
  Arms: CD patient with CO2 insufflation; UC patient with CO2 insufflation

SUMMARY:
Patients with inflammatory bowel disease (IBD) frequently undergo endoscopic examination and may suffer from diagnostic procedures. Independent from IBD patients, colonoscopy is usually performed using air insufflation, however recent data indicates a superior role of carbon dioxide (CO2) as an insufflation gas during colonoscopy. Using CO2 leads to a lower degree of patient's discomfort. The role of CO2 as an insufflation gas for colonoscopy in IBD patients remains undetermined, wherefore this study aims to address this issue.

DETAILED DESCRIPTION:
Patients with inflammatory bowel disease (IBD) suffer from a chronic inflammatory course of disease. To stage the course of disease endoscopic procedures including colonoscopy may be required and especially IBD patients with their inflamed gut may suffer from repetitive endoscopic examinations including colonoscopy. Independent from IBD patients, colonoscopy is usually performed using air insufflation, however recent data indicates a superior role of carbon dioxide (CO2) as an insufflation gas during colonoscopy. Using CO2 leads to a lower degree of patient's discomfort which has been mainly demonstrated in groups of patients undergoing cancer surveillance colonoscopies and who do not suffer from IBD. Therefore the role of CO2 as an insufflation gas for colonoscopy in IBD patients remains undetermined and this study aims to address this issue. For pain assessment a visual analogue scale will be used. As the primary outcome measure, the investigators will compare the differences in pain level 1h after colonoscopy (comparison of carbon dioxide to air insufflation). For the secondary outcome measure the investigators will compare the differences in pain level 3h, 6h and 24h after colonoscopy (comparison of carbon dioxide to air insufflation).

ELIGIBILITY:
Inclusion Criteria:

* Patient with inflammatory bowel disease
* Indication for colonoscopy
* Age 18-80 years
* signed consent form

Exclusion Criteria:

* Consent form not signed
* Age < 18 or above 80 yrs
* Pregnancy or Breast-Feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2017-09-03 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of colonoscopy related abdominal pain 1 hour after examination assessed by a visual analogue pain scale in patients with inflammatory bowel disease | Pain level assessment 1 hour after colonoscopy
  For pain assessment a visual analogue scale will be used. For the primary outcome measure, the investigators will compare the difference in pain level 1 hour after colonoscopy (comparison of carbon dioxide to air insufflation).

SECONDARY OUTCOMES:
Comparison of colonoscopy related abdominal pain 3 hours, 6 hours and 24 hours after examination assessed by a visual analogue pain scale in patients with inflammatory bowel disease | Pain level assessment 3 hours, 6 hours and 24 hours colonoscopy
  For pain assessment a visual analogue scale will be used. For the secondary outcome measure, the investigators will compare the differences in pain level 3 hours, 6 hours and 24 hours after colonoscopy (comparison of carbon dioxide to air insufflation).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lenze, MD, Principal Investigator — Department of Medicine B, University Hospital Muenster
Locations (1):
- Unversity Clinic Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided